CLINICAL TRIAL: NCT05908318
Title: Preoperative Olfactory Training Reduces the Incidence of Postoperative Delirium in Elderly Patients Undergoingorthopedic Surgeries: a Prospective Randomized Controlled Clinical Study
Brief Title: Effect of Preoperative Olfactory Training on Postoperative Delirium in the Elderly Undergoing Orthopedic Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SYSKY-2023-137-02
Record Dates: First submitted 2023-05-29; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Preoperative Olfactory Training; Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Olfactory Training

STUDY DESIGN:
Intervention Model Description: Recruited patients will be randomly divided into control group and olfactory training group.The olfactory training group was performed 24-48h before surgery used phenylethyl alcohol (rose), phytol (press tree), citronella (lemon), eugenol (clove) 4 kinds of smell，twice a day for three days.
Who Masked: Outcomes Assessor
Masking Description: In this study, different researchers will be responsible for randomization, olfactory training, anesthesia and visit. Due to the peroperative olfactory training in the olfactory training group, it is impossible to blind the participant and researchers implementing olfactory training.A researcher is responsible for assigning random numbers to ensure the randomness of the study groups. In order to ensure that the whole study is not affected by subjective factors, the researchers implementing and visiting are blinded, who do not know the anesthesia grouping, and are responsible for anesthsia, case enrollment screening, signing informed consent, preoperative and postoperative delirium evaluation, postoperative pain evaluation, complications and safety evaluation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group conducts standard preoperative preparation
- olfactory training group (Experimental): The olfactory training group was performed 24-48h before surgery used phenylethyl alcohol (rose), phytol (press tree), citronella (lemon), eugenol (clove) 4 kinds of smell，twice a day for three days.
  Interventions: Behavioral: olfactory training

INTERVENTIONS:
Behavioral: olfactory training — In this group, patients were performed 24-48h before surgery used phenylethyl alcohol (rose), phytol (press tree), citronella (lemon), eugenol (clove) 4 kinds of smell，twice a day for three days.
  Arms: olfactory training group

SUMMARY:
To observe whether preoperative olfactory training can reduces the incidence of postoperative delirium in elderly patients undergoing orthopedic surgeries, a prospective randomized controlled study method will be used in this study.

DETAILED DESCRIPTION:
450 elderly patients undergoing orthopedic surgeries (hip or knee replacement and laminectomy) under general anesthesia or combined spinal epidural anesthesia will be selected. They will be randomly divided into control group and olfactory training group.The olfactory training group was performed 24-48h before surgery used phenylethyl alcohol (rose), phytol (press tree), citronella (lemon), eugenol (clove) 4 kinds of smell，twice a day for three days. The general condition, operation, anesthesia and hospitalization related data of the patients will be recorded.

Outcome Measures： Incidence of postoperative delirium: The 3D-CAM scores of the control group and the olfactory training group were evaluated within 1-5 days after operation.

Degree of delirium：The MDAS of the control group and the olfactory training group were evaluated within 1-5 days after operation.

Pain：The VAS of the control group and the olfactory training group were evaluated within 1-5 days after operation.

Olfactory function：The TDI scores of the control group and the olfactory training group were evaluated in 3 days before operation and 48h after operation.

Cognitive function：The MoCA scores of the control group and the olfactory training group were evaluated in postoperative 5-7 days.

Markers: Delirium related markers and inflammatory factors in bloods was detected before surgery and after anesthesia. Delirium related markers and inflammatory factors in cerebrospinal fluid was detected after spinal puncture.

Subgroup analysis: patients were divided into delirium group and non-delirium group according to whether delirium occurred, and the data of the two groups were compared, including preoperative and postoperative olfactory function TDI scores, preoperative and postoperative VAS scores, nutritional scores, activity scores, and frailty index, Carlson comorbidity index, depression, anxiety state, sleep disturbance, etc., to screen risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoingorthopedic surgeries (hip or knee replacement and laminectomy) under general anesthesia or combined spinal-epidural anesthesia:
2. 65 years old ≤ age ≤ 90 years old, gender is not limited, ASA classification ≤ class III:
3. There is no recent history of surgery, and the operation time is ≥ 2 hours.
4. Able to communicate normally, able to cooperate and complete the cognitive function test. MMSE score >17.
5. Patients and their families are aware of and willing to participate.

Exclusion Criteria:

1. emergency surgery;
2. People with brain diseases or history of brain diseases such as cerebral infarction, stroke, etc.:
3. Have a history of neurological and psychological diseases, including Alzheimer's disease, Parkinson's, psychosis, etc.:
4. Illiteracy, severe hearing or visual impairment;
5. Those who have taken psychotropic drugs or abused psychotropic drugs within one month:
6. Sinusitis, previous nasal surgery history, nasal congestion, upper respiratory tract infection in the past two weeks, previously diagnosed rhinitis and other diseases that may affect olfactory function.
7. Patients who are allergic to pollen
8. Patients who cannot cooperate or refuse to sign informed consent

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | Postoperative 1-5 days
  The 3D-CAM scores

SECONDARY OUTCOMES:
Degree of delirium | Postoperative 1-5 days
  Memorial delirium assessment scale(MDSA)
Olfactory function | postoperative 48h compared to preoperative 72h
  The Sniffin' Sticks test involves testing odor for threshold and discrimination whilst blind folded and secondly odor identification. The sum of four odors responses ranges from 0-16. The sum of total score from odor Threshold, Discrimination and Identification (TDI) is a maximum of 48 points. The total score is graded as; normosmia equals or over 30.5 points, hyposmia 16.5-30 points and anosmia less than 16.5 points.
Cognitive function | postoperative 5-7 days
  Total score of the Montreal Cognitive Assessment (MoCA).
Postoperative pain | Postoperative 1-5 days
  Post-operative pain, measured in visual analogue scale (VAS),0:no pian, 10:worst pain.
Delirium related markers and inflammatory factors in bloods | immediate post-anesthesia compared to pre-operation
  These markers include:IL-6, IL-8, IL-10, TNF-α, IL-1β, CRP, N-terminal BNP, albumin, NSE, S-100B, Aβ-42 and T-tau, P-tau, S-100β
Delirium related markers and inflammatory factors in cerebrospinal fluid | immediate post-anesthesia compared to pre-operation
  These markers include:IL-6, IL-8, IL-10, TNF-α, IL-1β, albumin, NSE, S-100B, Aβ-42 and T-tau, P-tau, S-100β

IPD SHARING:
Plan to Share IPD: No